CLINICAL TRIAL: NCT04916821
Title: Investigation of Clinical Effectiveness of Propolis Extracts as Food Supplements in Patients With SARS-CoV-2(COVID-19)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trabzon Kanuni Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Betül Değer Kulaksız, assistant professor, Trabzon Kanuni Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00001
Record Dates: First submitted 2021-05-26; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Propolis

STUDY DESIGN:
Intervention Model Description: first group treated with water extracts of propolis second group treated with olive oil extracts of propolis including perga third group treated with no bee product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- water extract of propolis (Experimental): Patients given 2 ml of aqueous propolis extract (50mg / ml) orally 3 times a day for 1 week
  Interventions: Dietary Supplement: propolis
- olive oil extract of propolis including perga (Experimental): Patients given 1 ml oily propolis extract (64 mg / ml) + 1 ml oily perga extract (120 mg / ml) orally 3 times a day for 1 week
  Interventions: Dietary Supplement: propolis
- control (No Intervention): control group (patients not given any investigational product)

INTERVENTIONS:
Dietary Supplement: propolis — Propolis may be blocked virus entry to cells, and some receptor binding and some cell signal molecules
  Arms: olive oil extract of propolis including perga; water extract of propolis

SUMMARY:
Primary purpose: To investigate the effect of propolis, a food supplement product, on healing parameters in patients with COVID 19. Secondary purpose: To provide a new supportive treatment in Covid 19 treatment. In the present study to examine the effect of the use of propolis on healing parameters (laboratory and imaging) in patients with COVID 19; Propolis, which has antiviral properties, has also been used in humans in the COVID19 pandemic as of 2020. However, in these studies, an alcohol-soluble extract of propolis was used. Despite the disadvantages of its use in alcohol, it is clear that water and olive oil extracts of Propolis are safer for humans. Therefore, water extracts of propolis will be used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who do not need a ventilator who are inpatient in the Covid service
* Patients under the age of 60 who do not need a ventilator who are inpatient in the Covid service

Exclusion Criteria:

* patients do not have oral intake
* patients whose informed consent form is not approved
* patients who need a ventilator
* pregnant women
* children

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
radiological | Change from Baseline Lung Tomography Findings(Peripheral ground-glass opacities) at one week
  Lung tomography findings
laboratory parameters-2: ESR | Change from Baseline ESR findings at one week
  ESR
laboratory parameters-3: CRP | Change from Baseline CRP findings at one week
  CRP
laboratory parameters-4: D-Dimer | Change from Baseline D-Dimer findings at one week
  D-Dimer
laboratory parameters-5: Troponin | Change from Baseline Troponin findings at one week
  Troponin
laboratory parameters-6: sO2 | Change from Baseline sO2 findings at one week
  sO2
laboratory parameters-1: CBC | Change from Baseline CBC findings at one week
  CBC

CONTACTS AND LOCATIONS:
Overall Officials: Betül Değer Kulaksız, M.D, Study Chair — Trabzon Kanuni Education and Research Hospital
Locations (1):
- Trabzon Faculty of Medicine , Health Science University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Berretta AA, Silveira MAD, Condor Capcha JM, De Jong D. Propolis and its potential against SARS-CoV-2 infection mechanisms and COVID-19 disease: Running title: Propolis against SARS-CoV-2 infection and COVID-19. Biomed Pharmacother. 2020 Nov;131:110622. doi: 10.1016/j.biopha.2020.110622. Epub 2020 Aug 17. PMID 32890967
- [Background] Lima WG, Brito JCM, da Cruz Nizer WS. Bee products as a source of promising therapeutic and chemoprophylaxis strategies against COVID-19 (SARS-CoV-2). Phytother Res. 2021 Feb;35(2):743-750. doi: 10.1002/ptr.6872. Epub 2020 Sep 18. PMID 32945590